CLINICAL TRIAL: NCT02900027
Title: Placebo-Controlled, Dose-Escalation Study to Assess Safety, Tolerability, PK and PD of a GalNAc3 Conjugated Antisense Oligonucleotide Targeting ApoC-III, Administered Subcutaneously to Healthy Volunteers With Elevated Triglycerides
Brief Title: Safety, Tolerability, PK, and Pharmacodynamics(PD) of IONIS APOCIII-LRx in Healthy Volunteers With Elevated Triglycerides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IONIs-ApoCIII-LRx
Record Dates: First submitted 2016-08-23; First posted 2016-09-14 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Elevated Triglycerides (TG)
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IONIS-APOC-III-LRx (Experimental): Ascending single and multiple doses of IONIS-APOC-III-LRx by subcutaneous (SC) injection
  Interventions: Drug: Placebo Comparator
- Placebo (Normal Saline) (Placebo Comparator): Sterile Normal Saline (0.9% NaCl) calculated volume to match active comparator
  Interventions: Drug: APOC-III-L-Rx

INTERVENTIONS:
Drug: APOC-III-L-Rx — Ascending single and multiple doses of IONIS-APOC-III-LRx by subcutaneous (SC) injection
  Arms: Placebo (Normal Saline)
Drug: Placebo Comparator — Sterile Normal Saline (0.9% NaCl) calculated volume to match active comparator
  Arms: IONIS-APOC-III-LRx

SUMMARY:
The purpose is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of IONIS APOC-III-LRx given to healthy volunteer subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements
* Healthy males or females aged 18-65 inclusive
* Females must be non-pregnant and non-lactating, and either surgically sterile or post- menopausal
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method
* BMI < 35.0 kg/m2
* Subjects must have Fasting TG ≥ 90 mg/dL or ≥ 200 mg/dL depending on Cohort assignment

Exclusion Criteria:

* Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
* Treatment with another Study Drug, biological agent, or device within one-month of screening
* Regular excessive use of alcohol within 6 months of Screening
* Use of concomitant drugs unless authorized by the Sponsor Medical Monitor
* Smoking > 10 cigarettes a day
* Considered unsuitable for inclusion by the Principal Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple doses of IONIS- APOC-III-LRx - (incidence, severity, and dose-relationship of adverse effects and changes in the laboratory parameters) | Up to 183 days
  The safety and tolerability of IONIS- APOC-III-LRx will be assessed by determining the incidence, severity, and dose relationship of adverse effects and changes in the laboratory parameters by dose. Safety results in subjects dosed with IONIS APOC-III-LRx will be compared with those from subjects dosed with placebo.

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics of single and multiple doses of IONIS- APOC-III-LRx | Up to 183 days
  The maximum area under the curve (AUC) of IONIS- APOC-III-LRx will be assessed following single and multiple- dose SC administration
To evaluate the urine pharmacokinetics of single and multiple doses of IONIS¬-APOC-III-LRx | Up to 183 days
  The amount of IONIS-APOC-III-LRx excreted in urine at selected 24-hour intervals [Ae0-24h] will be determined.
To evaluate the plasma pharmacokinetics of single and multiple doses of IONIS- APOC-III-LRx | Up to 183 Days
  The maximum plasma concentration (Cmax) of IONIS- APOC-III-LRx will be assessed following single and multiple- dose SC administration
To evaluate the plasma pharmacokinetics of single and multiple doses of IONIS- APOC-III-LRx | Up to 183 days
  The maximum time to Cmax (Tmax) of IONIS- APOC-III-LRx will be assessed following single and multiple-dose SC administration

OTHER OUTCOMES:
Exploratory pharmacodynamic effects of IONIS-APOC-III-LRx | Up to 183 days
  Effects of IONIS-APOC-III-LRx on changes in levels of oxidized phospholipids associated with plasma apolipoprotein C-III (apoC-III) compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APOC-III-LRx | Up to 183 days
  Effects of IONIS-APOC-III-LRx on changes in levels of oxidized phospholipids associated with TG compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APOC-III-LRx | Up to 183 days
  Effects of IONIS-APOC-III-LRx on changes in levels of oxidized phospholipids associated with total cholesterol (TC) compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APOC-III-LRx | Up to 183 days
  Effects of IONIS-APOC-III-LRx on changes in levels of oxidized phospholipids associated with low density lipoprotein cholesterol (LDL-C) compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APOC-III-LRx | Up to 183 days
  Effects of IONIS-APOC-III-LRx on changes in levels of oxidized phospholipids associated with high density lipoprotein cholesterol (HDL-C) compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APOC-III-LRx | Up to 183 days
  Effects of IONIS-APOC-III-LRx on changes in levels of oxidized phospholipids associated with non-high density lipoprotein cholesterol (non-HDL-C) compared to baseline.
Exploratory pharmacodynamic effects of IONIS-APOC-III-LRx | Up to 183 days
  Effects of IONIS-APOC-III-LRx on changes in levels of oxidized phospholipids associated with very low density lipoprotein cholesterol (VLDL-C) compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Faulknor, Principal Investigator — BioPharma Services
Locations (1):
- BioPharma Services, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Alexander VJ, Xia S, Hurh E, Hughes SG, O'Dea L, Geary RS, Witztum JL, Tsimikas S. N-acetyl galactosamine-conjugated antisense drug to APOC3 mRNA, triglycerides and atherogenic lipoprotein levels. Eur Heart J. 2019 Sep 1;40(33):2785-2796. doi: 10.1093/eurheartj/ehz209. PMID 31329855